CLINICAL TRIAL: NCT01147445
Title: Phase I Study to Determine the Safety and Immunogenicity of an Oral ETEC Candidate Vaccine, Attenuated, Recombinant Double Mutant Heat-Labile Toxin (dmLT) From Enterotoxigenic Escherichia Coli
Brief Title: Phase I Study of ETEC Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0066
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2012-06-25

CONDITIONS: Gastroenteritis Escherichia Coli
Keywords: Enterotoxigenic Escherichia coli; vaccine
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1: 5 mcg dmLT (Experimental): 6 subjects to receive 5 micrograms (mcg) of dmLT vaccine.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 2: 25 mcg dmLT (Experimental): 6 subjects to receive 25 mcg of dmLT vaccine.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 3: 50 mcg dmLT (Experimental): 6 subjects to receive 50 mcg of dmLT vaccine.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 4: 100 mcg dmLT (Experimental): 6 subjects to receive 100 mcg of dmLT vaccine.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Cohort 5: 50 mcg or 100 mcg dmLT (Experimental): 12 subjects randomized, double-blinded, to receive either 50 mcg or 100 mcg of dmLT vaccine.
  Interventions: Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine

INTERVENTIONS:
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat labile enterotoxin. LT(R192G/L211A) is formulated as a freeze-dried (lyophilized), white to off-white cake, containing 700 micrograms of vaccine protein in a 3 mL, multi-dose, Wheaton Serum Vial. Vaccine dosage levels: 5, 25, 50, 100 micrograms as a single, oral dose.

SUMMARY:
The purpose of this study is to learn if a new candidate vaccine (dmLT) against ETEC (E. coli infection) is safe. This vaccine will be tested to see what effects it has on the body and the ability of the vaccine to help the body resist disease. Researchers want to find the highest dose of dmLT vaccine that can be given without causing severe side effects. Most E. coli bacteria are harmless to humans and can even be beneficial. However, some are harmful, and can cause diarrhea. About 32 healthy adults, ages 18-45, will participate in this study. This study will require volunteers to stay in the research facility for several nights. Participants will be assigned to receive 1 of 4 vaccine doses by mouth. Study procedures include: stool samples, blood samples, and documenting side effects. Participants will be involved in study related procedures for about 8 months.

DETAILED DESCRIPTION:
Despite the public health burden of enterotoxigenic Escherichia (E.) coli (ETEC) on travelers, deployed soldiers and, most significantly, young children in the developing world, there is no licensed vaccine against ETEC enteritis. The rationale for using an E. coli heat labile enterotoxin (LT) (R192G/L211A) vaccine, also called double-mutant LT (dmLT), is that it is expected to be especially well tolerated by subjects. If dmLT is safe and immunogenic, it may become an anti-toxin vaccine or a component of other ETEC vaccine candidates, as well as an adjuvant for mucosal immunization. This is a phase I dose escalation study, in which 4 cohorts of 6 subjects each will be enrolled and receive 5 micrograms (mcg), 25 mcg, 50 mcg, or 100 mcg of dmLT vaccine, plus a fifth cohort of 12 subjects which will be randomized and double-blinded to receive either 50 mcg or 100 mcg of dmLT vaccine. A Safety Monitoring Committee (SMC) will be convened for this study, and will review available safety data through the Day 8 visit for each cohort prior to making a recommendation to the Sponsor on whether or not to proceed to the next cohort. If a dose is not well tolerated as determined by the SMC review of the safety data, a Confirmation Cohort of 8 subjects will be enrolled and administered the previous dose. The first two cohorts will be enrolled simultaneously, dosed with investigational product, and observed to ensure the tolerability through Day 8 of the 5 mcg and 25 mcg dose levels. The first two cohorts will be dosed simultaneously based on the excellent safety record of these doses for the single mutant LT (LTR192G). Thereafter, dose escalation and subject enrollment will proceed in a step-wise fashion. Safety will be assessed by solicited symptoms/subject memory aid and laboratory evaluations. Adverse events (AE)s will be graded according to standardized criteria. The immunogenicity outcome measures of interest are the rate and titer of seroconversion with serum and fecal immunoglobulin A (IgA) anti-LT antibodies measured by ELISA and stimulation of anti-LT antibody secreting cells (ASC). The sample size was chosen based on the exploratory nature of this test article study that has not previously been given to humans. Participants will include 36 healthy adult male and female subjects, ages 18 to 45 inclusive. The primary objective of this study is to assess the safety of dmLT vaccine when administered as a single oral dose over a range of dose levels in healthy adult subjects. The primary objective of Cohort 5 will be to evaluate the safety and immunogenicity of the 50 µg and 100 µg doses of an orally administered dmLT vaccine in healthy adult subjects. The secondary objectives are to assess long-term safety follow-up from immunization through Month 6 post vaccination and to evaluate the immunogenicity of a single oral dose of dmLT vaccine over a range of doses in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

-Male or female ages 18-45, inclusive. -Provide written informed consent before initiation of any study procedures. -Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, and medication history. -Within 45 days of vaccination, have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), prothrombin time (PT), partial thromboplastin time (PTT), International Normalized Ratio (INR), C-reactive protein (CRP), and fibrinogen as defined in Appendix B. -Have normal screening laboratories for urine protein and urine glucose. -Demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination (passing grade is at least 70 percent). -Capable of understanding, consenting and complying with the entire study protocol including the inpatient period. -Female subjects must be of non-childbearing potential, (as defined as surgically sterile or postmenopausal for more than 1 year), or if of childbearing potential must be practicing abstinence or using an effective licensed method of birth control (e.g., history of hysterectomy or tubal ligation; use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), cervical sponges, diaphragms, condoms with spermicidal agents, or must have a vasectomized partner) within 2 months of vaccination and must agree to continue such precautions during the study and for 30 days after the Day 28 study visit. Male subjects must agree not to father a child for 90 days after the Day 0 study visit. A woman is eligible if she is monogamous with a vasectomized male. -Agrees not to participate in another clinical trial during the study period. -Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine.

Exclusion Criteria:

-Women who are pregnant or lactating or have a positive serum pregnancy test at screening or positive urine pregnancy test upon admission to inpatient facility. -Abnormal Vital signs, defined as: Hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days; or (heart rate <55 at rest on 2 separate days) Respiratory rate >17 -Temperature >/= 38.0 C (100.4 F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days of administration of dmLT. -Active positive Hepatitis B, C, and Human Immunodeficiency Virus (HIV) serologies. -Have a positive urine drug screen. -Subjects who are unwilling or unable to cease smoking for the duration of the inpatient stay. -History of antimicrobial treatment in the 2 weeks before ingestion of dmLT. -Received previous experimental E. coli, LT, or cholera vaccines or live E. coli or Vibrio cholerae challenges; or previous infection with cholera or diarrheagenic E. coli. -Abnormal bowel habits as defined by fewer than 3 stools per week or more than 2 stools per day in the past 6 months. -History of chronic gastrointestinal illness, including severe dyspepsia (mild or moderate heartburn or epigastric pain occurring no more than 3 times per week is permitted), lactose intolerance, or other significant gastrointestinal tract disease. -Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy. -History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy. -Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed). -Have a diagnosis of schizophrenia or other major psychiatric diagnosis. -Receiving the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, molindone, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. NOTE: Subjects who are receiving a single antidepressant drug and are stable for at least 3 months before enrollment without de-compensating symptoms, will be allowed to be enrolled in the study. -History of receiving immunoglobulin or other blood product within the 3 months before enrollment in this study. -Traveled to certain Enterotoxigenic Escherichia coli (ETEC) endemic areas within the past 3 years or raised in a cholera or ETEC endemic area. -Received any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before enrollment in this study. -An acute or chronic medical condition that, in the opinion of the investigator, would render ingestion of dmLT unsafe or would interfere with the evaluation of responses. This includes, but is not limited to: known or suspected immunodeficiency, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, history of diabetes, cancer (other than a healed skin lesion), heart disease (in the hospital for a heart attack, history of irregular heart beat or fainting caused by an irregular heart beat), unconsciousness (other than a single brief "concussion"), seizures (other than with fever when subject was a child <5 years old), asthma requiring treatment with inhaler or medication in the prior 2 years, autoimmune disease or eating disorder, and transpla nt recipients. -Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study. -History of alcohol or drug abuse in the last 5 years. -Planned to travel outside of the USA in the time between vaccination and 28 days following the vaccination. -Unable to spend 4 days as an inpatient. -Any condition that would, in the opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol. -Use of prescription and over-the-counter (OTC) medications that contain acetaminophen, aspirin, ibuprofen, and other nonsteroidal anti-inflammatory drugs within 48 hours prior to receiving the investigational product. -Use of prescription acid suppression medication or OTC antacids within 72 hours of investigational product administration. -Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation. -Subjects who plan to travel to an ETEC endemic area during the long-term safety follow-up period (6 months) of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2012-06-08 (Actual); Study Completion 2012-06-08 (Actual)

PRIMARY OUTCOMES:
Safety of double-mutant E. coli heat labile enterotoxin (dmLT) vaccine. The occurrence of dose escalation halting events. Additional safety includes the incidence and severity of adverse events (AEs) and changes in laboratory and clinical parameters. | Day 0, follow-up clinic visits (Days 8 ±1, 14 ±2, 28 ±2), and months 2 ±2 weeks, 6 ±2 weeks, by telephone. After Day 28 post vaccination, adverse event follow-up limited to only SAEs, non-routine medical visits, and new-onset chronic medical conditions.

SECONDARY OUTCOMES:
Adverse Events. | Through 6 months.
Immunogenicity: stimulation of anti-dmLT antibody secreting cells (ASC) measured by ELISPOT and seroconversion rates and geometric mean titers of serum anti-LT immunoglobulin (Ig) IgG and IgA antibodies and fecal anti-LT IgA antibodies measured by ELISA. | Serum and stool collected on Days 8, 14, and 28.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center - Gastroenterology, Hepatology and Nutrition, Cincinnati, Ohio

REFERENCES:
- [Background] El-Kamary SS, Cohen MB, Bourgeois AL, Van De Verg L, Bauers N, Reymann M, Pasetti MF, Chen WH. Safety and immunogenicity of a single oral dose of recombinant double mutant heat-labile toxin derived from enterotoxigenic Escherichia coli. Clin Vaccine Immunol. 2013 Nov;20(11):1764-70. doi: 10.1128/CVI.00464-13. Epub 2013 Sep 18. PMID 24049109